CLINICAL TRIAL: NCT05596136
Title: Artery Alert - Revolutionizing the Diagnosis of Peripheral Arterial Disease
Brief Title: Novel Blood Biomarker for Peripheral Arterial Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Unity Health Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Mohammad Qadura, Principal Investigator; Surgeon-Scientist, Division of Vascular Surgery, Department of Surgery, Unity Health Toronto
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 2-Unity
Record Dates: First submitted 2022-10-04; First posted 2022-10-27 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Artery Alert — A device for the measurement of the protein of interest that can be administered in a physician's office without requiring any capital equipment

SUMMARY:
This study focuses on validating the clinical efficacy of a novel point of care diagnostic blood test for peripheral arterial disease (PAD) within a large, heterogeneous patient population. With support from CIHR, our aim is to overcome the knowledge-to-action gaps regarding inadequate and underutilized diagnostic modalities in patients with PAD who at high risk of cardiovascular (CV) events. We propose to ascertain the diagnostic accuracy of a blood-based marker for PAD by cross-validating it with the current gold-standard.

DETAILED DESCRIPTION:
Lower extremity peripheral arterial disease (PAD) is a common presentation of atherosclerosis, affecting 256 million people globally. Despite its prevalence, approximately 50% of PAD patients are either undiagnosed, misdiagnosed, or get diagnosed late in their disease status4. Asymptomatic patients, in particular, account for these devastatingly high rates of under-diagnosis. Studies demonstrate that over 60% of PAD patients are asymptomatic, and their paucity of clinical symptoms makes diagnosis immensely difficult. Concerningly, asymptomatic PAD patients are at a similar risk of death, heart attacks and limb loss as clinically symptomatic PAD patients.

Consequently, PAD patients (both symptomatic and asymptomatic) receive delayed treatment subsequently face a higher risk of lower extremity amputation, CV events, and mortality. A possible solution to reduce the incidence of PAD induced morbidity and mortality is through early diagnosis, as studies have shown that it leads to improved survival and limb salvage rates16. However, diagnosing patients with PAD in its early stages is a major challenge faced by many physicians today, due to the limitations associated with the current PAD diagnostic modalities.

Currently, the diagnosis of PAD is established through physical exam, clinical history, and arterial imaging including the ankle brachial index (ABI) - the ratio of the brachial artery blood pressure to the ankle blood pressure. This test serves as the only validated screening tool for PAD and an ABI of ≤0.90 has a 75% sensitivity and 86% specificity. However, the ABI is challenging to use within primary care practice for a few reasons. First, it is not a fully reliable diagnostic tool for PAD. For instance, 25% of diabetic patients have falsely elevated ABI values due to incompressible calcified vessels. Second, since the majority of PAD patients are asymptomatic (60%), primary care physicians rarely refer them for an ABI test for screening. Third, the ABI has geographical limitations as well, as it is only conducted at specialized centers and is not widely available at all clinics. This is particularly true in rural areas and in Indigenous communities - thus compromising health equity.

To validate the challenges physician face with using the ABI as a screening test for PAD, we conducted customer interviews and a survey on 52 primary care physicians within Ontario. Our results confirm that primary care providers face several barriers with accessing and performing the ABI. These barriers include: the extensive training it requires, the length of time it takes in the physician's office (i.e. >15 minutes) and lack of access to specialized equipment (i.e. inaccessible). Furthermore, our data confirm that the ABI measurement is under-utilized and often incorrectly performed within primary care practice - complimenting previously published findings in the literature. Most notably, physicians surveyed in our study were extremely enthusiastic about the potential of a novel blood test for diagnosing PAD. They remarked a blood test that can be ordered/administered during annual physical examinations for patients with cardiovascular risk factors will prove useful in identifying and caring for asymptomatic PAD patients in particular and triaging them to appropriate early vascular care.

Based on the unmet need identified in the survey, our research team discovered, patented, and validated, a novel blood-based biomarker of PAD. In this study, we aim to ascertain the diagnostic accuracy of a blood-based marker for PAD by cross-validating it with the current gold-standard (ABI).

ELIGIBILITY:
Inclusion Criteria:

* Male or female (sex)
* At least 40 years or older
* Willingness to comply with study protocol and provide written informed consent

Exclusion Criteria:

* Stage 4 and 5 renal failure according to the Kidney Disease Outcomes Quality Initiative clinical guidelines
* Inability to provide informed consent
* Acute/recent diagnosis (within past 3 months) of acute coronary syndrome, as defined by the American College of Cardiology

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 548 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Number of patients that Artery Alert correctly diagnoses with PAD by cross validating with the current gold standard | 4 years